CLINICAL TRIAL: NCT06876805
Title: The Role of Contrast Enhanced Ultrasond (Ceus), in the Characterization of Focal Liver Lesions Indeterminate to Second-level Methods
Brief Title: The Role of Ceus in the Characterization of Focal Liver Lesions Indeterminate to Second-level Methods
Acronym: InFoLIL
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: InFoLIL
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Focal Liver Lesion
Keywords: CEUS; Ultrasound; Liver; HCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with focal liver lesions indeterminated at II level imaging methods
  Interventions: Diagnostic Test: CEUS or Contrast enhanced Ultrasound

INTERVENTIONS:
Diagnostic Test: CEUS or Contrast enhanced Ultrasound — CEUS performed as normal clinical practice
  Other Names: Contrast enhanced ultrasound

SUMMARY:
The primary objective of the study is to determine the accuracy of CEUS in characterizing (as benign or malignant) focal liver lesions for which CT, MRI and/or PET have not been conclusive.

DETAILED DESCRIPTION:
The study conducted will be a non-profit, observational, non-pharmacological, cross-sectional, but also partly cohort, retrospective and prospective study. The study is cross-sectional in nature, but will require 6 months of follow-up to evaluate the gold standard reference outcome in patients diagnosed with a benign pathology that does not require further investigations, and in patients with suspected malignant lesion for which histological diagnosis has not been performed on biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* CEUS performed performed in the last 6 months a CT, MRI and/or PET not decisive in characterizing a liver lesion.
* Obtaining informed consent.

Exclusion Criteria:

* Technical impossibility to perform the ultrasound evaluation.
* Documented allergy to the ultrasound contrast medium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have previously resulted positive to CT, MRI and/or PET scans for liver lesions but with no information on the nature of the lesion and that will undero CEUS for further characterization of the lesion(s) will be consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
CEUS diagnostic accuracy | 2 years
  CEUS diagnostic accuracy in determining the nature of focal liver lesions

CONTACTS AND LOCATIONS:
Overall Officials: Carla Serra, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Policlinico Sant'Orsola Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided